CLINICAL TRIAL: NCT07398989
Title: A Clinical Study to Assess Efficacy and Tolerability of a Topical Skincare Product on Adults With Mature, Crepey Skin
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GLI.04.US.SL.048
Record Dates: First submitted 2026-01-13; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-10

CONDITIONS: Crepey Skin; Aging Skin; Photo-aged Skin
MeSH Terms: interventions — cetyl alcohol, propylene glycol, sodium lauryl sulfate non-lipid cleansing lotion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Skincare Product Treatment (Experimental): Subjects will apply topical skincare products to the body.
  Interventions: Drug: Cetaphil

INTERVENTIONS:
Drug: Cetaphil — Subjects will apply Cetaphil Hydrating and Firming Cream Skin Activator to the knees, thighs, hands, and all of the body at least twice daily. Subjects will use Cetaphil Daily Facial Moisturizer SPF 35 as needed.

SUMMARY:
Subjects having mild-to-moderate crepiness, photodamage, and loss of firmness will apply a topical skincare regimen to the knees, thighs, hands, and all over the body. Evaluations of the regimen's efficacy will be conducted at 4 weeks, 8 weeks, and 12 weeks post-baseline.

ELIGIBILITY:
Inclusion Criteria:

1. Adult subjects aged 40-60 years
2. Females and males
3. Any Fitzpatrick skin types (FST) I-VI, with effort to include minimum n = 2 for each category per Site
4. Any races, with effort to include minimum 10% minority (n = 3 for both Sites) such as American Indian or Alaska Native, Eastern/Southeastern Asian, South Asians, Black or African American, Native Hawaiian or Other Pacific Islander.
5. Any ethnicities, with effort to include minimum 10% (n = 3 for both Sites) of Hispanic, Latino, or Spanish origin.
6. History of skin fragility and prone to bruising, i.e., dermatoporosis.
7. Having mild-to-moderate (score 3-6 according to a modified Griffiths scale, where 0 = none and 9 = severe) score for the following parameters on the knees and lower thighs: crepiness, photodamage, firmness
8. Subjects in general good health
9. Willing to stop using current topical skincare products for the duration of the study.
10. Willing to replace current skincare products with study product for the duration of the study.
11. Willing to have investigational areas photographed, i.e., knees, lower thighs, hands.
12. Willing to change into clinic-provided clothes for study photography of the knees/lower thighs.
13. For biopsy subgroup (n = 5) at Site 1: having healthy immune system, willing to have skin biopsies on the upper knees
14. For all subjects at Site 2: willing to undergo bruise induction procedure on the upper knees
15. For female subjects of childbearing potential, she must not be pregnant, breastfeeding or planning pregnancy during the course of the study. Subjects must be willing to take a urine pregnancy test (UPT) prior to study start. Females of non-childbearing potential, e.g., post-menopausal, hysterectomy, or bilateral ovariectomy, are not required to have a UPT.
16. Ability to read, understand, and give consent for participation in the study.
17. Willing to sign a photography release.
18. Agreement to comply with all the time commitments and adhere to the procedural requirements of the protocol, and to report to the Site on the day(s) and at the time(s) scheduled for the assessments.

Exclusion Criteria:

* Pregnant, breastfeeding, or planning pregnancy during the course of the study. 2. Subject with any known allergies or hypersensitivity to any cosmetics, personal care products, and/or fragrances. 3. History of cancer within the past 5 years 4. History or presence of any skin condition/dermatologic disease on the test areas (knees, lower thighs, hands) that might interfere with the evaluation of study parameters and/or put the subject at significant risk (according to the Investigator's judgment) if the subject takes part to the trial. 5. Planning on having surgeries and/or invasive medical procedures during the course of the study. 6. For biopsy subgroup at Site 1 and all subjects at Site 2:

  1. History of allergy or hypersensitivity to anesthetics or lidocaine
  2. Have been diagnosed with a bleeding disorder
  3. Have experienced excessive bleeding after other medical procedures
  4. Currently taking blood-thinning medications (e.g., aspirin, aspirin-containing medications, warfarin or heparin), immunosuppressive medications or systemic steroids.
  5. History of keloid formation or hypertrophic scarring 7. Having clinically active bacterial, fungal, or viral skin infections or those who have a history of skin infections. 8. The subject has received, applied, or ingested the following treatments within the specified time frame prior to the Baseline visit:

  <!-- -->

  1. Oral isotretinoin (Accutane) or other oral retinoids - 6 months.
  2. Avita, Differin, Renova, Retin-A, Retin-A Micro, Soriatane, or Tazorac - 3 months.
  3. Prescription-strength skin-lightening products for the test areas (e.g., hydroquinone, tretinoin, alpha/beta/poly-hydroxy acids, 4-hydroxyanisole alone or in combination with tretinoin, etc.) - 3 months.
  4. Over-the-counter (OTC) retinol-containing products (with retinaldehyde, retinyl palmitate, retinyl esters, retinyl acetate, or retinyl propionate, etc.) - 4 weeks.
  5. Other OTC anti-wrinkle, skin-lightening, or other product or topical or systemic products known to affect skin aging or dyschromia (eg, products containing alpha/beta/poly-hydroxy acids, emblica extract, Gigawhite, hydroquinone, lemon juice extract [topically], Q-10, soy, systemic or licorice extract [topically], Tego® Cosmo C250, vitamin C[topically]) - 2 weeks.
  6. Antibiotics (except penicillin) - 4 weeks
  7. Benzoyl peroxide, azelaic acid, zinc, corticosteroids, other topical treatments (including laser) - 2 weeks
  8. Corticosteroids (except inhaled corticosteroids or intrathecal corticosteroids) - 4 weeks
  9. Immunomodulators, including biologics - 6 months
  10. Non-steroidal anti-inflammatory drugs - 2 weeks 9. Having observable sunburn, suntan, scars, nevi, excessive hair, tattoos, piercings, or other dermal conditions on the test areas that might interfere with the trial results in the opinion of the Investigator. 10. Planning intense UV exposure during the study (i.e., occupational exposure to the sun, sunbathing, tanning salon use, phototherapy, etc.). 11. Having clinically significant abnormality according to the Investigator during enrollment. 12. Having any disease that might interfere with the trial results in the opinion of the Investigator. 13. Current smokers of tobacco products. 14. Unwilling to refrain from use of prohibited medication during the clinical trial. 15. Other condition preventing the subject from entering the study in the Investigator's opinion, (e.g., subjects failing baseline assessments, subjects not likely to avoid other cosmetic treatments in the treatment area, subjects anticipated to be unavailable or incapable of understanding the study assessments or having unrealistic expectations of the treatment result). 16. The subject is currently participating in any other clinical trial of a drug or device OR past participation in any other clinical trial within the 30 days prior of Screening. 17. Study site personnel, close relatives of the study site personnel (e.g., parents, children, siblings, or spouse), or employees and close relatives of employees at the Sponsor company.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-12 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Change of clinical grading compared to baseline | Baseline, Week 4, Week 8, Week 12
  Clinical grading of efficacy parameters will be performed at both study sites. The efficacy parameters will be assessed by the Investigators at the knees and lower thighs using a modified Griffiths' 10-point scale , with 0 indicating best possible condition and 9 indicating worst possible condition. Half-point scores may be used as necessary to more accurately describe the skin condition. A decrease in scores indicates an improvement.
Change in skin hydration as measured by Corneometer | Baseline, Week 4, Week 8, Week 12
  Corneometer (Courage + Khazaka, Germany) measurements will be taken in triplicate to assess skin hydration. The Corneometer measures in Corneometer units from 0 (no water at all) - 120 (on water). Measurements will be taken on the lower thigh/upper knee at 9 locations. An increase in scores indicates an improvement.
Change in tolerability grading compared to baseline | Baseline, Week 4, Week 8, Week 12
  Tolerability assessment will be evaluated at both study sites. The areas for evaluation on the body are knees and lower thighs. Investigator will assess erythema, edema, and dryness using a 4-point analog scale (with half-point scores used as necessary to better describe the clinical condition). A score of 0 indicates best possible condition, and a score of 3 indicates worst possible condition.
Change in skin quality measured by macroscopic imaging (Visioscan) | Baseline, Week 4, Week 8, Week 12
  Macroscopic imaging procedure of skin texture will be performed using Visioscan® VC 20plus on all subjects, at Site 1 only. Images will be taken of each subject's upper knee (left or right). Imaging location will be the same at each timepoint.
Measured pH values consistent with baseline | Baseline, Week 4, Week 8, Week 12
  Skin pH measurements will be performed using pH Meter on all subjects, at Site 1 only. Triplicate measurements will be taken on the upper knee (left or right). pH value will be expressed in two decimals. A lack of significant change in values indicates maintenance of skin pH.

OTHER OUTCOMES:
Visual change in bruising intensity compared to baseline | Baseline, Week 12
  Bruise induction procedure will be performed on all subjects at Site 2 only. At Baseline and D84/W12, subjects will participate in a cupping procedure after all assessments are completed to induce bruising. Bruising intensity will be visually assessed on the Bruise Visibility Scale, which is a 1-5 scale, with 1 indicating the bruise is barely visible, and 5 indicating the bruise is prominently or unmistakably visible. A decrease in scores indicates an improvement.
Change in bruising duration compared to baseline bruise induction | Baseline, Week 12
  Bruise induction procedure will be performed on all subjects at Site 2 only. At Baseline and D84/W12, subjects will participate in a cupping procedure after all assessments are completed to induce bruising. Subjects will capture photos of the bruises daily until bruise resolution. A decrease in bruise duration indicates an improvement in bruise resolution.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Ablon Skin Institute & Research Center, Manhattan Beach, California
  - Clinical Research Center of the Carolinas, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No